CLINICAL TRIAL: NCT05816967
Title: Rationalisation of Polypharmacy by the RASP-instrument (Rationalisation of Home Medication by an Adjusted STOPP-list and Discharge Counselling of Geriatric Inpatients: a Prospective, Clinical Trial
Brief Title: Rationalisation of Polypharmacy by the RASP-instrument and Discharge Counselling of Geriatric Inpatients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Interference with other trials on the same ward
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S59694
Record Dates: First submitted 2022-05-24; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Polypharmacy
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): In the monocentric interventional part of the study, the effect of discharge counseling on the acceptance of pharmacotherapeutic recommendations will be evaluated 1 and 3 months after discharge.
  Interventions: Procedure: Medication review and discharge counseling

INTERVENTIONS:
Procedure: Medication review and discharge counseling — Medication reconciliation of home therapy will be performed by the clinical pharmacist through a standardized form. Next, the clinical pharmacist will perform a medication review, based on but not limited to the RASP list (Van der Linden 2014). The goal is optimization of therapy. Before discharge the clinical pharmacist will perform a second medication review, together with the treating physician and a medication reconciliation in orde to provide the best possible discharge medication list. The medication list will be provided 3 times: once for the patient and/or his/her caregiver, once for the general practitioner and once for the primary care pharmacist. Finally the clinical pharmacist will have a counseling session with the patient and/or his/her caregiver.

SUMMARY:
Systematic evaluation of polypharmacy in geriatric patients, through a validated list by a clinical pharmacist. The goal is reduction of potentially inappropriate medications (PIMs). A brief counseling session with the patient and/or his/her caregiver will be part of the intervention.

DETAILED DESCRIPTION:
This project is focused on the systematic evaluation of polypharmacy in older patients admitted to the acute geriatric wards of a university hospital. Polypharmacy will be identified through a validated list by a clinical pharmacist. The goal is reduction of potentially inappropriate medications (PIMs). Before hospital discharge the hospital pharmacist will have a brief counseling session with the patient and/or his/her caregiver in order to discuss the medication list and to enhance compliance.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the patient and/or his/her caregiver
* Admission through the emergency department of patients coming from home or a residential care facility

Exclusion Criteria:

* Patients not speaking Dutch
* Patients admitted for end of life care
* Patients not taking any drugs on admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Acceptance rate of the pharmacotherapeutic recommendations, provided by the clinical pharmacist by the general practitioner. | 1 month (30 days) after discharge
  Acceptance rate of the pharmacotherapeutic recommendations, provided by the clinical pharmacist by the general practitioner.
Acceptance rate of the pharmacotherapeutic recommendations, provided by the clinical pharmacist by the general practitioner. | 3 month (90 days) after discharge
  Acceptance rate of the pharmacotherapeutic recommendations, provided by the clinical pharmacist by the general practitioner.

SECONDARY OUTCOMES:
Number of drug intakes at discharge versus at admission. | At discharge from the index hospitalization (as mentioned in the discharge medication scheme) vs on admission (during the first 72 hours of the index hospitalization)
  Number of drug intakes at discharge versus at admission.
Number of drugs at discharge versus at admission. | At discharge from the index hospitalization (as mentioned in the discharge medication scheme) vs on admission (during the first 72 hours of the index hospitalization)
  Number of drugs at discharge versus at admission.
Number of drugs adapted by the treating physician based on recommendations by the clinical pharmacist that are not included in the RASP list. | At discharge from the index hospitalization (as mentioned in the discharge medication scheme), compared to the medication list obtained on admission (this is, during the first 72 hours of the hospitalization)
  Number of drugs adapted by the treating physician based on recommendations by the clinical pharmacist that are not included in the RASP list.
Difference in number of potentially inappropriate medications identified through the RASP list on admission versus at discharge | At discharge from the index hospitalisation (as mentioned in the discharge medication scheme) versus on admission (medication list obtained in the first 72 hours) of the index hospitalization
  Difference in number of potentially inappropriate medications identified through the RASP list on admission versus at discharge
Number of potentially inappropriate medications on admission, at discharge and at the follow-up moments (1 and 3 months after discharge) | On admission (medication list obtained in the first 72 hours of the admission), at discharge (as mentioned in the discharge medication scheme), 1 (30 days) month after discharge, 3 months (90 days) after discharge
  Number of potentially inappropriate medications on admission, at discharge and at the follow-up moments (1 and 3 months after discharge)
Mortality during admission | During the index hospitalization, from admission to the emergency ward until moment of death on the geriatric ward, assessed up to 72 hours after death.
  Mortality during admission
Number of falls during hospitalization | During the index hospitalization, from admission on the emergency ward until discharge from the geriatric ward, assessed within 72 hours after discharge.
  Number of falls during hospitalization
Number of fractures during hospitalization | during the index hospitalization, from admission to the emergency ward until discharge from the geriatric ward, assessed within 72 hours after discharge.
  Number of fractures during hospitalization
Length of stay | During the index hospitalization, from admission to the emergency ward until discharge from the geriatric ward, assessed within 72 hours after discharge.
  Length of stay
Readmission rate 3 months after discharge | 3 months (90 days) after discharge from the geriatric ward (index hospitalization), assessed at day 90
  Readmission rate 3 months after discharge
Number of fractures at 3 months after discharge | 3 months (90 days) after discharge from the geriatric ward (index hospitalization), assessed at day 90
  Number of fractures at 3 months after discharge
Number of falls 3 months after discharge | 3 months (90 days) after discharge from the geriatric ward (index hospitalization), assessed at day 90
  Number of falls 3 months after discharge
Mortality at 3 months after discharge | 3 months (90 days) after discharge from the geriatric ward (index hospitalization), assessed at day 90
  Mortality at 3 months after discharge
Category of potentially inappropriate medications identified through the RASP list on admission and at discharge | On admission (medication list obtained in the first 72 hours of the admission), at discharge (as mentioned in the discharge medication scheme)
  Category of potentially inappropriate medications identified through the RASP list on admission and at discharge
Category of drugs adapted by the treating physician based on recommendations by the clinical pharmacist that are not included in the RASP list. | During the course of the index hospitalization, defined as the period between discharge from the geriatric ward and admission to the geriatric department. The outcome parameter will be assessed within 72 hours of discharge.
  Category of drugs adapted by the treating physician based on recommendations by the clinical pharmacist that are not included in the RASP list.
Number of drugs at follow-up (1 month and 3 months after discharge) | 1 month (30 days) and 3 months (90 days) after the index hospitalization
  Number of drugs at follow-up (1 month and 3 months after discharge)
Number of drug intakes at follow-up (1 month and 3 months after discharge) | 1 month (30 days) and 3 months (90 days) after the index hospitalization
  Number of drug intakes at follow-up (1 month and 3 months after discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hias, Pharm D, Principal Investigator — UZ Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No